CLINICAL TRIAL: NCT05090163
Title: Prep Plus: Supporting Upper Limb Practice in Community Dwelling Stroke Survivors
Brief Title: Prep Plus: Upper Limb Stroke Rehabilitation in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Northern Ireland Chest Heart and Stroke (Other)
Responsible Party: Principal Investigator, Katy Pedlow, Dr Katy Pedlow, Principal Investigator, University of Ulster
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21/NI/0043
Record Dates: First submitted 2021-09-22; First posted 2021-10-22 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: Upper limb; Physical activity; Rehabilitation
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Intervention Model Description: Each site will deliver 6 weeks of the intervention / control with a new set of participants before post intervention qualitative measures are used to inform the design of the next wave.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREP group (Active Comparator): Control group
  Interventions: Other: PREP
- PREP Plus group (Experimental): Intervention group
  Interventions: Other: PREP Plus

INTERVENTIONS:
Other: PREP Plus — Group based exercise in addition to PREP exercises
  Arms: PREP Plus group
Other: PREP — Group based exercise
  Arms: PREP group

SUMMARY:
PREP Plus aims to create support for those who have survived stroke(s) and are still experiencing weakness in the upper limbs. In conjunction with the PREP programme, and based on the GRASP programme, the aim is to evaluate the feasibility, acceptability, and efficacy of an upper limb intervention support for survivors. Integration of an evidence based upper limb programme to an established physical activity programme will be a feasible method to support long term upper limb rehabilitation to community dwelling stroke survivors.

DETAILED DESCRIPTION:
The main objectives for overall study is to assess acceptability of the demand of the trial as well as the PREP Plus intervention placed on survivors and their carers. Within this mixed methods study, the investigators aim to recruit participants in a total of three waves. Each site will deliver 6 weeks of the intervention / control with a new set of participants before post intervention qualitative measures (focus groups and 1:1 interviews) are used to inform the design of the next wave. With having the trial in three waves, their objective is to optimise the design of upper limb rehab and the delivery by therapists with preparing them with adequate training and resources aimed toward upper limb rehab in survivors of stroke.

Participant recruitment will integrate into the current PREP programme design.

All participants will complete one hour of circuit-based exercises followed by one hour of education. The exercise stations will focus on lower body/cardiovascular fitness station and upper limb strength exercises. Each week the amount of time spent at each station will be increased by 30 seconds resulting in a final 3 minutes at each station. Those in the intervention group, will have an additional five exercises that focus on upper limb stretching, arm stretching, hand stretching, coordination, and hand skills.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of stroke

Have completed statutory rehabilitation

Able to follow two part written or spoken commands

Are medically fit to complete exercise, as determined by their GP

Having an impairment of their upper limb, as identified by the participant and/ or their community stroke team.

Exclusion Criteria:

Pain score of 5/more in their impaired upper limb. Not participating in any other trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Rating of Everyday Arm-use in the Community and Home (REACH) Scale: Measuring change in upper limb use from baseline to 6 weeks | 6 weeks
  upper limb use

SECONDARY OUTCOMES:
Edinburgh Warwick Questionnaire: Measuring change in mental wellbeing from baseline to 6 weeks | 6 weeks
  Mental wellbeing and quality of life measure
10 meter walk test: Measuring change in walking speed from baseline to 6 weeks | 6 weeks
  functional performance measure
Timed Get up and Go [TUG] test: Measuring change in lower limb function from baseline to 6 weeks | 6 weeks
  lower limb functional performance test

OTHER OUTCOMES:
Focus group with participants | end of 6 weeks
  Overall experience: Stroke survivor experience
1:1 interviews with intervention therapist | end of 6 weeks
  Determine optimum design considering acceptability, practicality and resources. Therapist experience and practicality of delivery
Caregivers questionnaire provided at post intervention. | end of 6 weeks
  Overall experience: View accessibility of the group from a carer point of view
Recruitment log | Throughout the study completion, an average of 1 year
  Recruitment rate: Percentage of eligible participants approached and agreed to participate Refusal reason: Participant reason for refusal linked to (A) Study process, (B) Intervention
Weekly attendance records | Throughout the study completion, an average of 1 year
  Retention rates: Percentage of participants who completed the 6 week programme

CONTACTS AND LOCATIONS:
Overall Officials: Katy Pedlow, Principal Investigator — Ulster University
Locations (1):
- Ulster University, Jordanstown, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Any published data from the study will be available on the Ulster University data repository
Supporting Information: Study Protocol
Time Frame: September 2023
URL: https://pure.ulster.ac.uk/en/persons/katy-pedlow

REFERENCES:
- [Background] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Background] Veerbeek JM, van Wegen E, van Peppen R, van der Wees PJ, Hendriks E, Rietberg M, Kwakkel G. What is the evidence for physical therapy poststroke? A systematic review and meta-analysis. PLoS One. 2014 Feb 4;9(2):e87987. doi: 10.1371/journal.pone.0087987. eCollection 2014. PMID 24505342
- [Background] Rand D, Eng JJ. Predicting daily use of the affected upper extremity 1 year after stroke. J Stroke Cerebrovasc Dis. 2015 Feb;24(2):274-83. doi: 10.1016/j.jstrokecerebrovasdis.2014.07.039. Epub 2014 Dec 18. PMID 25533758
- [Background] Pollock A, St George B, Fenton M, Firkins L. Top 10 research priorities relating to life after stroke--consensus from stroke survivors, caregivers, and health professionals. Int J Stroke. 2014 Apr;9(3):313-20. doi: 10.1111/j.1747-4949.2012.00942.x. Epub 2012 Dec 11. PMID 23227818
- [Background] Kwah LK, Harvey LA, Diong J, Herbert RD. Models containing age and NIHSS predict recovery of ambulation and upper limb function six months after stroke: an observational study. J Physiother. 2013 Sep;59(3):189-97. doi: 10.1016/S1836-9553(13)70183-8. PMID 23896334
- [Background] Taub E, Uswatte G, Mark VW, Morris DM. The learned nonuse phenomenon: implications for rehabilitation. Eura Medicophys. 2006 Sep;42(3):241-56. PMID 17039223
- [Background] Pang MY, Harris JE, Eng JJ. A community-based upper-extremity group exercise program improves motor function and performance of functional activities in chronic stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2006 Jan;87(1):1-9. doi: 10.1016/j.apmr.2005.08.113. PMID 16401430
- [Background] Rand D, Eng JJ. Disparity between functional recovery and daily use of the upper and lower extremities during subacute stroke rehabilitation. Neurorehabil Neural Repair. 2012 Jan;26(1):76-84. doi: 10.1177/1545968311408918. Epub 2011 Jun 21. PMID 21693771
- [Background] Arwert H, Schut S, Boiten J, Vliet Vlieland T, Meesters J. Patient reported outcomes of hand function three years after stroke. Top Stroke Rehabil. 2018 Jan;25(1):13-19. doi: 10.1080/10749357.2017.1385232. Epub 2017 Oct 12. PMID 29025365
- [Derived] Pedlow K, Kennedy NC, Klempel N, Eng JJ, Adamson G, Hylands J, Hughes N, Campbell Z, McDonough S. Post-rehabilitation programme to support upper limb recovery in community-dwelling stroke survivors: a mixed methods cluster-feasibility controlled trial. BMJ Open. 2024 Oct 15;14(10):e088301. doi: 10.1136/bmjopen-2024-088301. PMID 39414298
- [Derived] Pedlow K, McDonough S, Klempel N, Hylands J, Hughes N, Campbell Z, Eng JJ, Stephenson A, Kennedy N. PREP Plus combined postrehabilitation programme to support upper limb recovery in community-dwelling stroke survivors: protocol for a mixed-methods, cluster-assigned feasibility study. BMJ Open. 2023 Jan 20;13(1):e069016. doi: 10.1136/bmjopen-2022-069016. PMID 36669847
- See also: Global Health Estimates — https://www.who.int/data/global-health-estimates
- See also: Stroke Guidelines — https://www.rcplondon.ac.uk/guidelines-policy/stroke-guidelines